CLINICAL TRIAL: NCT06645249
Title: Multicenter, Randomized Clinical Trial to Evaluate the Cardioverter Capacity of Amiodarone Pre-electrical Cardioversion in Persistent Atrial Fibrillation
Brief Title: Evaluation of Cardioverter Capacity of Amiodarone Pre-electrical Cardioversion in Persistent Atrial Fibrillation
Acronym: PERIVERSION
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Institut Investigacio Sanitaria Pere Virgili (Other)
Collaborators: Spanish Society of Cardiology (Other); Sociedad Espanola de Cardiologia (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-507201-34-00; SCC 2023 (Other Grant/Funding Number: Societat Catalana de Cardiologia); SEC/FEC-INV-CLI 23/24 (Other Grant/Funding Number: Sociedad Española de Cardiologia); 2023-507201-34-00 (EU CTIS Number)
Record Dates: First submitted 2024-09-30; First posted 2024-10-16 (Actual); Last update posted 2024-12-02 (Actual); Status verified 2024-11

CONDITIONS: Atrial Fibrillation (AF)
Keywords: Atrial fibrillation; Electrical cardioversion; amiodarone; Pharmacological cardioversion
MeSH Terms: conditions — Atrial Fibrillation | interventions — Amiodarone; Anti-Arrhythmia Agents

STUDY DESIGN:
Intervention Model Description: This is a multicenter randomized phase IV open clinical trial. Patients with persistent AF (≥7 days duration) electively referred for CVE will be selected.
  Two amiodarone regimens administered pre-CVE will be compared evaluating their cardioverter efficacy. Patients will be randomized to 2 groups:
  c. Treatment impregnation with amiodarone starting one month before ECV (600 mg/day 1st week, 400 mg/day 2nd week and 200 mg/day thereafter until ECV).
  d.Treatment impregnation with amiodarone 800 mg/day started 5 days before ECV.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Amiodarone orally impregnation starting one month before ECV (Experimental): Treatment impregnation with amiodarone starting one month before ECV (600 mg/day 1st week, 400 mg/day 2nd week and 200 mg/day thereafter until ECV).
  Interventions: Drug: Amiodarone (Antiarrhythmic drug)
- Amiodarone orally impregnation started 5 days before ECV (Active Comparator): Treatment impregnation with amiodarone 800 mg/day started 5 days before ECV.
  Interventions: Drug: Amiodarone (Antiarrhythmic drug)

INTERVENTIONS:
Drug: Amiodarone (Antiarrhythmic drug) — Comparing 2 regimes of amiodarone pre-electrical cardioversion witn ECG monitoring

SUMMARY:
Phase: IV Population: Sample size= 122 patients; male and female; ≥ 18 y.o.; patients with persistent atrial fibrillation referred for electrical cardioversion; performed in Spain Number of Sites: 4 Study Duration: 15/10/2024 - 15/5/2026 Subject Participation Duration: 2-4 months (depending on the arm) Description of Agent or Intervention: amiodarone

Objectives:

Primary: To compare the efficacy of amiodarone in pre-ECV reversal to sinus rhythm in a one-month impregnation regimen versus a 5-day regimen Secondary: 1) Identify days from initiation of pre-ECV amiodarone to reversion to SR using a mobile device paired to the mobile phone; 2) To compare the joint efficacy in the reversion to SR pre-ECV and in the maintenance of SR at 1 month after ECV of a one-month pre-ECV amiodarone impregnation regimen vs a 5-day regimen

Description of Study Design: Multicenter randomized open clinical trial. 122 Patients with persistent AF (≥7 days duration) electively referred for CVE will be included. Two amiodarone regimens administered pre-CVE will be compared evaluating their cardioverter efficacy. Patients will be randomized to 2 groups:

1. Treatment impregnation with amiodarone starting one month before ECV (600 mg/day 1st week, 400 mg/day 2nd week and 200 mg/day thereafter until ECV).
2. Treatment impregnation with amiodarone 800 mg/day started 5 days before ECV. Estimated Time to Complete Enrollment: 13 months

DETAILED DESCRIPTION:
4.3 RISK AND BENEFITS (if any) The study will compare two peri-ECV AAD regimens of amiodarone in the range of those recommended in the technical data sheet and label (16). For this reason, the risks of participation in the study would be equivalent to those present in standard clinical practice.

5. OBJECTIVES AND ENDPOINTS 5.1 OBJECTIVES: 5.1.1 Primary Objective i. To compare the efficacy of amiodarone in pre-ECV reversal to sinus rhythm in a one-month impregnation regimen versus a 5-day regimen 5.1.2 Secondary Objectives i. Identify days from initiation of pre-ECV amiodarone to reversion to SR using a mobile device paired to the mobile phone.

ii. To compare the joint efficacy in the reversion to SR pre-ECV and in the maintenance of SR at 1 month after ECV of a one-month pre-ECV amiodarone impregnation regimen vs a 5-day regimen 5.2 ENDPOINTS 5.2.1 Endpoint (s) for the primary objective i. Reversal to sinus rhythm pre-ECV (number of patients) 5.2.2 Endpoint (s) for the secondary objectives i. Days until reversal to sinus rhythm ii. Maintenance of sinus rhythm at 1 month after cardioversion 5.3 HYPOTHESIS:

1. In patients with persistent AF referred to ECV, a long amiodarone impregnation regimen (one month pre-CVE) would induce pharmacological cardioversion in about a fifth of patients and would be superior to a short impregnation regimen (5 days).
2. Reversal to SR induced by the administration of pre-CVE amiodarone may occur in a vulnerable period for embolic events in patients in whom OAC is initiated pre-CVE. The use of a device that monitors the ECG daily will be useful to know when the reversion to pre-CVE RS occurs.
3. The proportion of patients who maintain the SR at one month post-CVE will be similar in a long regimen vs. a short regimen of pre-CVE amiodarone.

6. STUDY DESIGN This is a multicenter randomized phase IV open clinical trial. Patients with persistent AF (≥7 days duration) electively referred for CVE will be selected. After verifying that they meet the inclusion and exclusion criteria, candidates will be invited to participate in the study. Patients will receive information about the study and those who agree to participate will sign the informed consent.

Two amiodarone regimens administered pre-CVE will be compared evaluating their cardioverter efficacy. Patients will be randomized to 2 groups:

c. Treatment impregnation with amiodarone starting one month before ECV (600 mg/day 1st week, 400 mg/day 2nd week and 200 mg/day thereafter until ECV).

d. Treatment impregnation with amiodarone 800 mg/day started 5 days before ECV. Patients who do not revert to SR pre-ECV will be treated with ECV. Those who have pharmacologically reverted to SR or who have had a successful CVE will be treated with amiodarone 200 mg/day after restoration of SR. A one-month follow-up will be carried post-ECV to evaluate the maintenance of SR. ECV will be carried out as per standard clinical practice with 200 J biphasic energy and, if ineffective, maximum energy will be used.

According to the ESC clinical practice guidelines for AF, adequate anticoagulation is a necessary requirement for at least 3 weeks before ECV to avoid the risk of embolism associated with cardioversion. Patients on chronic anticoagulation will be started on the assigned pre-ECV amiodarone regimen after inclusion. Patients who are not already receiving anticoagulant treatment will begin anticoagulant treatment with direct anticoagulants. In this case, they will wait 3 weeks before starting the amiodarone regimen to avoid the risk of embolism during this period.

At baseline visit, the patient will be given a mobile electrocardiographic monitoring device to determine which patients revert to SR and the time of reversal. Patients will record a daily pre-ECV ECG strip that will be transmitted to the investigator team of each participating center. During the post-ECV follow-up month, patients will send a weekly ECG via the mobile monitoring device. During clinical visits a physical examination, ECG, vital signs, blood samples collection, record of concomitant medication and collection of adverse events will be performed.

No other AADs (except beta-blockers or calcium antagonists) will be allowed during the study. Patients who experience recurrence of AF or adverse side effects will be discontinued from the study.

ELIGIBILITY:
Inclusion Criteria:

1. Patients ≥18 years old.
2. Persistent atrial fibrillation (≥ 7 days duration).
3. Referred for elective electrical cardioversion.
4. Signing of the informed consent

Exclusion Criteria:

1. Need of urgent electrical cardioversion
2. Mean Heart rate <50 bpm
3. Planned ablation < 1 month after ECV.
4. Treatment with anti-arrhythmic drugs (IC, III) the last 7 days previous to inclusion (in the case of amiodarone on the 30 days previous to inclusion)
5. Atrial fibrillation post-cardiac surgery
6. New York Heart Association (NYHA) Class IV heart failure
7. Left ventricular ejection fraction (LVEF) ≤30%
8. History of thyroid disease (hyperthyroidism or hypothyroidism)
9. Known hepatobiliary disease (acute hepatitis, cirrhosis...) or ALT/AST > 3 x upper limit of normal (ULN)
10. Allergy, intolerance, or known hypersensitivity to study medication
11. Women of childbearing potential unwilling to use contraceptive measures
12. Participation in another clinical trial involving investigational drugs
13. Life expectancy less than 12 months
14. Rheumatic mitral stenosis of any degree or severe mitral or aortic valve dysfunction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 122 (Estimated)
Dates: Start 2024-12-10 (Estimated); Primary Completion 2026-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
Reversal to sinus rhythm pre-electrical cardioversion | From date of enrollment until the date of electrical cardioversion, up to 8 weeks
  Number of patients who revert to sinus rhythm before electrical cardioversion

SECONDARY OUTCOMES:
Days until reversal to sinus rhythm | From date of enrollment until date of electrical cardioversion, up to 8 weeks
  Number of days from enrollment to reversion to sinus rhythm
Maintenance of sinus rhythm at 1 month after cardioversion | From date of reversion to sinus rhythm until 1 month later
  Number of patients who remain in sinus rhythm at 1 month after reversion to sinus rhythm (pharmacological or electrical)

CONTACTS AND LOCATIONS:
Locations (4):
- Spain (4):
  - Hospital Universitari Germans Trias i Pujol, Badalona
  - Hospital de la Santa Creu i Sant Pau, Barcelona
  - Hospital Universitari de Sant Joan, Reus
  - Hospital Clínico Universitario de Santiago, Santiago de Compostela

IPD SHARING:
Plan to Share IPD: Yes
After requirement, IPD (without data who allow identify a subject) could be shared with other investigators.